CLINICAL TRIAL: NCT02707640
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of the Safety and Tolerability of N-Acetylcysteine in Patients With Idiopathic Pulmonary Fibrosis With Background Treatment of Pirfenidone
Brief Title: A Study to Assess the Safety and Tolerability of N-Acetylcysteine When Administered With Pirfenidone to Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA29976; 2012-000564-14 (EudraCT Number)
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Acetylcysteine; pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo; Drug: Pirfenidone
- N-Acetylcysteine (Experimental)
  Interventions: Drug: N-acetylcysteine; Drug: Pirfenidone
- Pirfenidone (Other): Background therapy
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Matching Placebo — Matching Placebo, oral administration, three times daily for 24 weeks.
  Arms: Matching Placebo
Drug: N-acetylcysteine — N-acetylcysteine, 600 mg, oral administration, three times daily for 24 weeks.
  Arms: N-Acetylcysteine
Drug: Pirfenidone — Pirfenidone, at least 1602 mg/day, oral administration, for 32 weeks, during the wash-out and screening period and for at least 8 weeks prior to randomization.

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled safety and tolerability study of N-acetylcysteine or placebo in participants with mild to moderate idiopathic pulmonary fibrosis (IPF) receiving background pirfenidone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms consistent with IPF of >=3 months' duration (relative to Day 1)
* Must have been on a dose of pirfenidone not less than 1602 mg/day for at least 8 weeks prior to randomization at Day 1
* Able to understand the importance of adherence to study treatment and the study protocol and willing to follow all study requirements, including the concomitant medication restrictions, throughout the study
* Women of childbearing capacity were required to have a negative serum pregnancy test before treatment and must have agreed to maintain highly effective contraception by practicing abstinence or by using at least two methods of birth control from the date of consent through the end of the study
* Diagnosis of usual interstitial pneumonia (UIP) or IPF by high-resolution computed tomography (HRCT) and surgical lung biopsy. Previous HRCT scans, typically and if available, one at the point of time of diagnosis and one more recent, made during the last year before study inclusion, will be used and assessed by a central Reading Committee

Exclusion Criteria:

* Significant clinical worsening of IPF between screening and Day 1 of study, in the opinion of the investigator
* Unlikely to comply with the requirements of this study, in the opinion of the investigator
* Patient-reported cigarette smoking within 3 months of screening or unwilling to avoid use of tobacco products throughout the study
* History of clinically significant environmental exposure known to cause pulmonary fibrosis (PF), including but not limited to drugs (such as amiodarone), asbestos, beryllium, radiation, and domestic birds
* Known cause of interstitial lung disease, including but not limited to radiation, drug toxicity, sarcoidosis, hypersensitivity pneumonitis, and cryptogenic organizing pneumonia
* Clinical diagnosis of any connective tissue disease, including but not limited to scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus, and rheumatoid arthritis
* Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis, urinary tract infection, or cellulitis (as a diffuse inflammation of connective tissue and or skin)
* Any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next 6 months (relative to Day 1). This does not include minor surgical procedures for localized cancer (e.g., basal cell carcinoma, squamous skin carcinoma)
* History of severe hepatic impairment or end-stage liver disease
* History of end-stage renal disease requiring dialysis
* History of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous 6 months (relative to Day 1)
* Any condition that, in the opinion of the investigator, may have been significantly exacerbated by the known side effects associated with the administration of N-acetylcysteine taken as a single medication
* Suspected intolerance, allergy, or hypersensitivity to pirfenidone or any of its components
* Known intolerance, allergy, or hypersensitivity to N-acetylcysteine or any of its components

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (65):
- Austria (3):
  - Graz
  - Innsbruck
  - Salzburg
- Belgium (3):
  - Brussels
  - Leuven
  - Mont-godinne
- Denmark (3):
  - Aarhus
  - Hellerup
  - Odense C
- France (12):
  - Bobigny
  - Brest
  - Bron
  - Dijon
  - Lille
  - Marseille
  - Montpellier
  - Paris
  - Reims
  - Rennes
  - Toulouse
  - Tours
- Germany (20):
  - Bad Berka
  - Bamberg
  - Berlin
  - Bochum
  - Bonn
  - Coswig
  - Donaustauf
  - Essen
  - Freiburg im Breisgau
  - Giessen
  - Greifswald
  - Hamburg
  - Heidelberg
  - Immenhausen
  - Magdeburg
  - Marburg
  - München
  - Münnerstadt
  - Solingen
  - Würzburg
- Italy (11):
  - Napoli, Campania
  - Cattinara Trieste, Friuli Venezia Giulia
  - Trieste, Friuli Venezia Giulia
  - Rome, Lazio
  - Catania, Liguria
  - Milan, Lombardy
  - Monza, Lombardy
  - Orbassano, Piedmont
  - Pisa, Tuscany
  - Siena, Tuscany
  - Padua, Veneto
- Sweden (4):
  - Falun
  - Lund
  - Stokholm, Solna
  - Uppsala
- United Kingdom (9):
  - Bristol
  - Cambridge
  - Exeter
  - Leeds
  - Liverpool
  - London
  - Oxford
  - Sheffield
  - Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetylcysteine (NAC): Participants randomized to this arm were administered 600 milligram (mg) NAC orally three times daily and a dose of pirfenidone of at least 1602 mg/day for 24 weeks. Participants were to be on a dose of pirfenidone of at least 1602 mg/day for a minimum of 8 weeks prior to randomization and were followed until 4 weeks after last study treatment dose.
- Placebo: Participants randomized to this arm were administered matching placebo orally three times daily and a dose of pirfenidone of at least 1602 mg/day for 24 weeks. Participants were to be on a dose of pirfenidone of at least 1602 mg/day for a minimum of 8 weeks prior to randomization and were followed until 4 weeks after last study treatment dose.
Period: Overall Study
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Started | 61 | 62
Completed | 52 | 55
Not Completed | 9 | 7
Not completed — Adverse Event | 4 | 2
Not completed — Death | 1 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Participant's Personal Decision | 1 | 2
Not completed — Sponsor Discretion | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all participants who were consented, were randomized, and received at least 1 dose of double-blind study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine (NAC) | Placebo | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (7.99) | 67.5 (6.22) | 67.1 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 53 | 51 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Reductions
Description: Percentage of participants with dose reductions in N-Acetylcysteine and placebo cohorts during the 24-week treatment period.
Time Frame: From baseline up to 24 weeks
Population: mITT population included participants who received at least 1 dose of double-blind study medication (NAC or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 60 | 62
percentage of participants | 5 | 4.8

2. Primary Outcome: Percentage of Participants With Early Treatment Discontinuations
Description: Percentage of participants with early treatment discontinuations in N-Acetylcysteine and placebo cohorts during the 24-week treatment period.
Time Frame: From baseline up to 24 weeks
Population: mITT population included participants who received at least 1 dose of double-blind study medication (NAC or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 60 | 62
percentage of participants | 14.8 | 11.3

3. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment.
Time Frame: Until 28 days from last dose of study treatment (Week 28)
Population: mITT Population included participants who received at least 1 dose of double-blind study medication (NAC or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 60 | 62
percentage of participants | 76.7 | 80.6

4. Primary Outcome: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, is life threatening, requires hospitalization or prolongation of hospitalization, or results in disability/incapacity, or congenital anomaly/birth defect.
Time Frame: Until 28 days from last dose of study treatment (Week 28)
Population: mITT population included who received at least 1 dose of double-blind study medication (NAC or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 60 | 62
percentage of participants | 5.0 | 6.5

5. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events Resulting in Permanent Discontinuation of Study Treatment
Time Frame: Until 28 days from last dose of study treatment (Week 28)
Population: mITT population included who received at least 1 dose of double-blind study medication (NAC or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 60 | 62
percentage of participants | 6.7 | 1.6

6. Primary Outcome: Percentage of Participants With Treatment-Emergent Deaths of All Causes
Time Frame: Until 28 days from last dose of study treatment (Week 28)
Population: mITT population included who received at least 1 dose of double-blind study medication (NAC or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 60 | 62
percentage of participants | 1.7 | 4.8

7. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events That Led to Dose Reduction or Temporary Discontinuation of Study Treatment
Time Frame: Until 28 days from last dose of study treatment (Week 28)
Population: mITT population included who received at least 1 dose of double-blind study medication (NAC or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 60 | 62
percentage of participants | 10 | 6.5

ADVERSE EVENTS:
Time Frame: Until 28 days from last dose of study treatment (Week 28)
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Serious Adverse Events (participants affected / at risk) | 3/60 | 4/62
Other Adverse Events (participants affected / at risk) | 46/60 | 50/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-Acetylcysteine (NAC) (N=60) | Placebo (N=62)
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
AORTIC ANEURYSM (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N-Acetylcysteine (NAC) (N=60) | Placebo (N=62)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 0
DIARRHOEA (Gastrointestinal disorders) | 6 | 9
NAUSEA (Gastrointestinal disorders) | 4 | 5
BRONCHITIS (Infections and infestations) | 4 | 3
INFLUENZA (Infections and infestations) | 3 | 1
NASOPHARYNGITIS (Infections and infestations) | 7 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1
HEADACHE (Nervous system disorders) | 1 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 4
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 8 | 1
RASH (Skin and subcutaneous tissue disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.